CLINICAL TRIAL: NCT04127799
Title: Northern Jiangsu Province People's Hospital
Brief Title: Integrative Management of Patients With Atrial Fibrillation Via Hospital-Community-Family-Based Telemedicine (HCFT-AF) Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Xiang Gu, Director of cardiology, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BL2019083
Record Dates: First submitted 2019-09-30; First posted 2019-10-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-02

CONDITIONS: Telemedicine; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital-Community-Family-Care Management Platform Online (Experimental): Hospital-Community-Family-Care Management Platform Online: the remote monitoring service platform on line based on community and family for subjects with CHF under the guidance of the regional central hospital
  Interventions: Other: Hospital-Community-Family-Care Management Platform Online; Other: Subjects with AF conventional treatment
- Subjects with AF conventional treatment (Active Comparator): Subjects with AF via conventional clinic visit according to the latest relevant guidelines
  Interventions: Other: Subjects with AF conventional treatment

INTERVENTIONS:
Other: Hospital-Community-Family-Care Management Platform Online — Subjects with Hospital-Community-Family-Care Management Platform online and those with the clinic follow up. In the program, participants were educated on the use of smart health-tracking devices and mobile application (APP) to collect and upload comprehensive data elements related to the risk of AF self-care management. They were also instructed to send text messages, view notifications, and receive individualized guidance on the mobile APP. The general practitioners viewed index of each participant on mobile APP and provided primary care periodically, and cardiologists in regional central hospital offered remote guidance and management if necessary. Outcomes assessed included accomplishments of the program, usability and satisfaction, engagement with the intervention, and changes of AF-related health behaviors.
  Arms: Hospital-Community-Family-Care Management Platform Online
Other: Subjects with AF conventional treatment — Subjects with standardized treatment according to latest guidelines via conventional visit.

SUMMARY:
Atrial fibrillation (AF) is one of the most common arrhythmias. Its repeated fluctuations in ventricular rate and irregular heart rhythm not only reduce exercise tolerance and quality of life, but also cause hemodynamic changes. The incidence of stroke is increased by 5 times or more compared with the average person. According to statistics, the annual mortality rate from stroke due to atrial fibrillation is about 20%-25%. Of course, like other cardiovascular diseases, atrial fibrillation occurs in a large proportion of the elderly population. According to statistics, 80% of patients with atrial fibrillation are 65 years of age or older. With the aging of the world's population, especially in the 21st century, the proportion of patients with atrial fibrillation has increased year by year. The treatment of atrial fibrillation involves many aspects such as switching to sinus rhythm, controlling heart rate and anticoagulant therapy, which is a long course affecting the adherence of AF patients. AF is a kind of disease that can be preventable and controllable. The out-of-hospital care for AF patients has been proved to reduce the mortality and unexpected readmission rate, but there are still high costs, poor compliance, low management efficiency and etc. Telemedicine was believed to solve these problems to further reduce the mortality of AF patients. The latest ESC Heart Failure Guidelines emphasis the significance of telemedicine in AF, however, it didn't provide a standardized AF remote management system.

DETAILED DESCRIPTION:
Subjects with Hospital-Community-Family-Care Management Platform online and those with the clinic follow up. In the program, participants were educated on the use of smart health-tracking devices and mobile application (APP) to collect and upload comprehensive data elements related to the risk of AF self-care management. They were also instructed to send text messages, view notifications, and receive individualized guidance on the mobile APP. The general practitioners viewed index of each participant on mobile APP and provided primary care periodically, and cardiologists in regional central hospital offered remote guidance and management if necessary. Outcomes assessed included accomplishments of the program, usability and satisfaction, engagement with the intervention, and changes of AF-related health behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Meeting the diagnostic criteria for atrial fibrillation;
3. Subjects can understand the situation of this study and agree to sign informed consent and continue to follow up.

Exclusion Criteria:

1. Atrial fibrillation caused by reversible causes, including: acute myocardial infarction (MI) within 1 month, acute myocarditis within 1 month, untreated hyperthyroidism, and electrophysiological examination, angiography, atrial fibrillation did not reappear after treatment;
2. There is no recurrence of atrial fibrillation after surgical treatment;
3. Due to other serious diseases, the expected survival time is less than 1 year;
4. Severe liver and kidney disease: serum creatinine>5.0mg/dl; ALT exceeds the reference value by more than 3 times (ALT> 100u/L);
5. Systolic or diastolic blood pressure ≥ 180/110mm Hg (1mm Hg = 0.133kPa), but can be selected after blood pressure control;
6. Diagnosed or suspected blood system diseases (except for mild to moderate anemia) leading to coagulopathy or accompanied by bleeding tendency;
7. Pregnant and lactating women;
8. Reluctance to use remote monitoring equipment (such as depression, dementia, impaired autonomy, lack of communication skills);
9. Participating in other treatment research or remote patient management programs;
10. The investigator consider that it is not suitable for joining the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of ischemic stroke | 1 year
The incidence of ischemic stroke | 2 year
Cardiovascular mortality | 1 year
Cardiovascular mortality | 2 year
all-cause mortality | 1 year
all-cause mortality | 2 year

SECONDARY OUTCOMES:
Incidence of systemic embolism | 2 year
  Systemic embolism (Limb, kidney, mesenteric artery, lung, retina, etc. must be confirmed by vascular ultrasound, angiography, surgery or biopsy)
Incidence of transient ischemic attack | 2 year
Incidence of severe hemorrhage | 2 year
  Fatal, life-threatening or potentially fatal bleeding requiring blood transfusion or surgical intervention
Incidence of slight hemorrhage | 2 year
  Obvious or recessive gastrointestinal bleeding, hemoptysis, nosebleeds, gross hematuria, subcutaneous congestion, anemia caused by blood loss, moderate chronic blood loss
Usability of the AF telemedicine platform intervention for patients | 4 months
  Perceived Health Web Site Usability Questionnaire (PHWSUQ)[1]
  1. Ease of finding specific information
  2. Ease of reading the information given
  3. Ease of listening to audio-information
  4. Overall appearance of the site
  5. Overall quality of graphics
  6. Quality of video information Ease-of-Use
  7. I found the use of this Web site easy to learn.
  8. Finding information on this Web site requires a lot of mental effort.
  9. Overall, I find this Web site is easy to use. Usefulness
  10. Using this Web site will help me understand specific health problem(s).
  11. Using this Web site will help me improve my knowledge about health.
  12. Using this Web site will help me maintain better health habits. Strongly disagree 1 2 3 4 5 6 7 Strongly agree For each independent assignment, a higher score means a better outcome.
Changes of lifestyles and healthy behaviors | 4 months
  Patients lifestyles and behaviors, associated with the occurrence and progress of AF, were collected at baseline, and 4 months through interviews, with the purpose of evaluating changes in self-management of patients.
Drug adherence | 4 months
  Patients drug adherence was assessed via the Pharmacy Quality Alliance adherence measure at baseline and 4 months individually.
  Pharmacy Quality Alliance adherence measure
  1. I am convinced of the importance of my prescription medication
  2. I worry that my prescription medication will do more harm than good to me
  3. I feel financially burdened by my out-of-pocket expenses for my prescription medication Agree completely/ Agree mostly/ Agree somewhat/Disagree somewhat/ Disagree mostly/Disagree completely
  Note: Add up the total number of points from the checked boxes Score Interpretation 0: Low risk for adherence problems (>75% probability of adherence) 2-7: Medium risk for adherence problems (32-75% probability of adherence) 8+ High risk for adherence problems (<32% probability of adherence)
Engagement of the intervention | 4 months
  It was assessed objectively via daily Web portal log-ins and use of the mobile APP

CONTACTS AND LOCATIONS:
Overall Officials: Lei Sun, Master, Study Director — Department of cardiovascular medicine; Ye Zhu, Doctor, Principal Investigator — Department of cardiovascular medicine; Xiaolin Sun, Doctor, Principal Investigator — Department of cardiovascular medicine; Jiang Jiang, Master, Principal Investigator — Department of cardiovascular medicine
Locations (1):
- Department of cardiovascular medicine,Northern Jiangsu Hospital, Yangzhou, Jiangsu, China

REFERENCES:
- [Derived] Jiang J, Gu X, Cheng CD, Li HX, Sun XL, Duan RY, Zhu Y, Sun L, Chen FK, Bao ZY, Zhang Y, Shen JH. The Hospital-Community-Family-Based Telemedicine (HCFT-AF) Program for Integrative Management of Patients With Atrial Fibrillation: Pilot Feasibility Study. JMIR Mhealth Uhealth. 2020 Oct 21;8(10):e22137. doi: 10.2196/22137. PMID 33084588